CLINICAL TRIAL: NCT05153655
Title: Safety and Tolerability of Local Ischemic Post-conditioning in Patients With Acute Ischemic Stroke After Mechanical Thrombectomy
Brief Title: Ischemic Post-conditioning in Acute Ischemic Stroke Thrombectomy
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTECT
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; ischemic postconditioning; endovascular thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ischemic post-conditioning group (Experimental): The safety and tolerability of ischemic post-conditioning will be investigated using 3+3 dose-escalation trial design.
  Interventions: Procedure: Local ischemic post-conditioning

INTERVENTIONS:
Procedure: Local ischemic post-conditioning — Direct local ischemic post-conditioning will be applied after successful recanalization of the culprit middle cerebral artery. Local ischemic post-conditioning consists of briefly repeated 4 cycles of occlusion and reperfusion (equal duration) of the initially occluded culprit middle cerebral artery using a balloon. The schedule of advancing duration is 0 " 1 " 2 " 3 " 4 " 5 min.

SUMMARY:
Ischemic post-conditioning is a neuroprotective strategy that has been proven to attenuate reperfusion injury in animal models of stroke. The purpose of this proof-of-concept study is to determine the safety and tolerability of ischemic post-conditioning in patients with acute ischemic stroke who are treated with mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;
* Acute ischemic stroke caused by middle cerebral artery M1 segment occlusion;
* Successful recanalization (mTICI 2b/3) after endovascular thrombectomy that confirmed by digital subtraction angiography;
* Written informed consent provided by the patients or their legal relatives.

Exclusion Criteria:

* Known diagnosis or clinical suspicion of cerebral vasculitis or fibromuscular dysplasia;
* Difficulty in reaching the designated position of the balloon used for ischemic post-conditioning;
* Stenting in the middle cerebral artery as rescue therapy during the thrombectomy procedures;
* > 2 times of balloon dilations as rescue therapy due to angioplasty during the thrombectomy procedures;
* Moderate or severe residual stenosis (≥ 50%) of the culprit artery after recanalization;
* Difficulty in complying with ischemic post-conditioning or other conditions that the investigator considered inappropriate for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with major response | Immediately after intervention on the day of ischemic post-conditioning
  Major response is any of the following:
  * Vessel perforation or rupture;
  * Reocclusion of the culprit vessel after post-conditioning;
  * Vessel dissection;
  * Severe vasospasm;
  * Ischemic post-conditioning related thrombotic events;
  * Rupture of the balloon used for post-conditioning.
  In the 3 + 3 design, 3 subjects are recruited for a given ischemic post-conditioning dose level. The trial is stopped if ≥ 2 of 3 subjects at a given dose level show major response. If only 1 of 3 subjects shows major response, 3 more subjects are recruited at a given dose level and a major response in any of them will stop the trial. Otherwise, same procedure is followed for the next ischemic post-conditioning dose level. Maximum tolerable dose will be the dose at the level before stopping of the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Related data will be shared if full study protocol and statistical analysis plan are provided with reasonable design.

REFERENCES:
- [Derived] Wu L, Wei M, Zhang B, Zhang B, Chen J, Wang S, Luo L, Liu S, Li S, Ren C, Hess DC, Song H, Zhao W, Ji X. Safety and Tolerability of Direct Ischemic Postconditioning Following Thrombectomy for Acute Ischemic Stroke. Stroke. 2023 Sep;54(9):2442-2445. doi: 10.1161/STROKEAHA.123.044060. Epub 2023 Jul 27. PMID 37497674
- [Derived] Wu L, Zhang B, Zhao W, Ji X, Wei M. Ischemic post-conditioning in acute ischemic stroke thrombectomy: A phase-I duration escalation study. Front Neurosci. 2022 Dec 8;16:1054823. doi: 10.3389/fnins.2022.1054823. eCollection 2022. PMID 36523440